CLINICAL TRIAL: NCT02940366
Title: the Long-term Effects of High-doSe pitavaStatin on Diabetogenicity in Comparison With Atorvastatin in Patients With Metabolic Syndrome (LESS-DM) Randomized Clinical Trial
Brief Title: Effect of High-dose Pitavastatin on Glucose Control in Patients With Metabolic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Hyung-Kwan Kim, Director, Division of Cardiology, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1406-027-584
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — pitavastatin; Atorvastatin

ARMS (2):
- Pitavastatin 4 mg orally daily (Experimental)
  Interventions: Drug: Pitavastatin 4 mg orally daily
- Atorvastatin 20 mg orally daily (Placebo Comparator)
  Interventions: Drug: Atorvastatin 20 mg orally daily

INTERVENTIONS:
Drug: Pitavastatin 4 mg orally daily — Pitavastatin 4 mg orally daily for 24months
  Arms: Pitavastatin 4 mg orally daily
Drug: Atorvastatin 20 mg orally daily — Atorvastatin 20 mg orally daily for 24months
  Arms: Atorvastatin 20 mg orally daily

SUMMARY:
This purpose of this study is to evaluate effect of high-dose Pitavastatin on glucose control in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as metabolic syndrome according to National cholesterol Education Program criteria
* Patients with hypercholesterolemia who required to start statin therapy

Exclusion Criteria:

* overt diabetes
* acute coronary syndrome within 2 months
* acute cerebrovascular event within 2 months
* recent treatment of statin within 1month
* recent diagnosed neoplasm
* recent diagnosed liver disease
* chronic kidney disease
* patients with myopathy
* pregnant women, nursing mothers, women with possibility of pregnant
* patients being adminstered cyclosporine
* patients with genetic disease such as galactose intolerance, lactose intolerance, glucose-galactose malabsorption
* patients with treatment cyclosporin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Absolute change in HbA1c level | baselina and after 24months treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park JB, Jung JH, Yoon YE, Kim HL, Lee SP, Kim HK, Kim YJ, Cho GY, Sohn DW. Long-term Effects of high-doSe pitavaStatin on Diabetogenicity in comparison with atorvastatin in patients with Metabolic syndrome (LESS-DM): study protocol for a randomized controlled trial. Trials. 2017 Oct 27;18(1):501. doi: 10.1186/s13063-017-2229-4. PMID 29078817